CLINICAL TRIAL: NCT02982993
Title: Hepatitis C Infection in World Trade Center Responders
Status: Completed | Type: Observational
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Collaborators: Centers for Disease Control and Prevention (U.S. Federal Agency); National Institute for Occupational Safety and Health (NIOSH/CDC) (U.S. Federal Agency)
Responsible Party: Sponsor
Other Study IDs: GCO 16-0912
Record Dates: First submitted 2016-12-02; First posted 2016-12-06 (Estimated); Last update posted 2019-02-04 (Actual); Status verified 2019-02

CONDITIONS: Hepatitis C Infection
Keywords: hepatitis C virus; linkage-to-care; World Trade Center Health Program cohort; Baby Boomer; risk factors for hepatitis C virus infection
MeSH Terms: conditions — Hepatitis C

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- WTC responders participating in HCV infection study: Members of the World Trade Center Health Program cohort born from 1945 to 1965 who choose to participate in this research study on hepatitis C infection

SUMMARY:
This study provides Hepatitis C virus screening to the members of the World Trade Center Health Program followed at the Icahn School of Medicine at Mount Sinai born during 1945-1965, and linkage to care for those found infected. The study will also determine if exposure to human remains, blood and/or bodily fluids during the World Trade Center Health Program activities are associated with Hepatitis C virus infection. These findings would be relevant to the larger United States population, especially to persons born during 1945-1965 who are at high risk of Hepatitis C virus infection.

DETAILED DESCRIPTION:
The purpose of the project is to determine if the World Trade Center Health Program cohort is at an increased risk of Hepatitis C virus infection, determine if human exposure to human remains, blood and/or body fluids during the World Trade Center recovery activities is associated with increased risk of Hepatitis C virus infection, and to determine if referral to a co-located site for Hepatitis C virus care is associated with improved linkage to Hepatitis C virus care in the members of the World Trade Center Health Program born during 1945 through 1965.

ELIGIBILITY:
Inclusion Criteria:

* Member of the World Trade Center Health Program at the Icahn School of Medicine at Mount Sinai
* Born during 1945-1965

Exclusion Criteria:

* None

Ages: 51 Years to 72 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The World Trade Center Health Program is a longitudinal cohort of World Trade Center rescue and recovery workers who participated in the World Trade Center Screening, Monitoring, and Treatment Program at the Icahn School of Medicine at Mount Sinai in New York, New York. Eligible World Trade Center responders were those who had worked or volunteered in lower Manhattan, or the Staten island landfill or barge-loading piers for 4 hours or more from September 11, 2001, to September 14, 2001; 24 hours or more during September, 2001; 80 hours or more from September, 2001, to December, 2001. Persons enrolled in the World Trade Center Health Program and were born from 1945-1965 are eligible.
Sampling Method: Non-Probability Sample
Enrollment: 3906 (Actual)
Dates: Start 2016-12; Primary Completion 2018-07-12 (Actual); Study Completion 2018-07-12 (Actual)

PRIMARY OUTCOMES:
Prevalence of Hepatitis C virus infection | 2 years
  The investigator will measure the prevalence of Hepatitis C virus infection in 3900 World Trade Center Health program members to test the hypothesis that World Trade Center Health program members have an increased risk of Hepatitis C virus infection.

SECONDARY OUTCOMES:
Correlation between the exposure to human remains, blood and/or bodily fluids to hepatitis C virus infection. | 2 years
  The investigator will test the measure of association between exposure to human remains, blood and / or bodily fluids and risk of hepatitis C virus infection, while adjusting for type of activity during work at World Trade Center site and use of personal protective equipment.

CONTACTS AND LOCATIONS:
Overall Officials: Stephanie H Factor, MD,MPH, Principal Investigator — Icahn School of Medicine at Mount Sinai; Paolo Bofetta, MD, MPH, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Icahn School of Medicine at Mount Sinai, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No